CLINICAL TRIAL: NCT06930274
Title: Stillbirth Risk Identification Using Multiparametric Ultrasound
Acronym: STIMULUS
Status: Recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Principal Investigator, Robert Rohling, Professor, University of British Columbia
Other Study IDs: H22-02803
Record Dates: First submitted 2025-04-01; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Perinatal Hypoxia
Keywords: Quantitative Ultrasound; Placenta; Stillbirth; Fetal Hypoxia
MeSH Terms: conditions — Stillbirth; Fetal Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — placenta
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to identify a novel biomarker for stillbirth.

Specifically the aim is to predict perinatal hypoxia using quantitative ultrasound from the placenta (QUS-P) between 35 and 37 weeks gestation.

DETAILED DESCRIPTION:
Funding: Wellcome Leap, In Utero Program

Primary outcome: Perinatal hypoxia

Background: Perinatal hypoxia is an inadequate supply to or utilization of oxygen by the fetus. It is typically diagnosed at delivery and can lead to serious medical complications, including encephalopathy, and ultimately stillbirth. Fetal hypoxia represents 23% of neonatal deaths worldwide.

Aim: To predict perinatal hypoxia using quantitative ultrasound from the placenta (QUS-P) between 35 weeks gestation and delivery.

Methods: Raw radio frequency data is collected during ultrasounds between 35 and 37 weeks gestation using ClariusTM (handheld ultrasound). All scans take place at BC Women's Hospital. QUS-P parameters are derived from the raw radio frequency data and analyzed using linear regression.

Impact: The ability to identify perinatal hypoxia as early as 35 weeks gestation will allow for additional monitoring as well as efforts to prepare for immediate intervention if necessary (e.g. c-section, resuscitation, neonatal cooling), prevent progression to encephalopathy, and ultimately stillbirth.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant with singleton
2. Age 19 years or older
3. Provision of informed consent
4. Planning to deliver at BC Women's Hospital
5. 38 weeks gestation or less

Exclusion Criteria:

1. Pregnant with multiples
2. Not planning to deliver at BC Women's Hospital
3. Less than 19 years of age
4. Greater than 38 weeks gestation

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential participants are recruited from the following sources:
  1. South Community Birth Program
  2. Maternal Fetal Medicine Clinics at BC Women's Hospital (EMMA and Fetal Monitoring)
Sampling Method: Non-Probability Sample
Enrollment: 282 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Presence of Perinatal Hypoxia at 35-37 weeks gestation | 35-37 weeks gestation
  Perinatal hypoxia is defined as meeting one or more of the following:
  1. Apgar < 7 at 5 minutes
  2. Umbilical artery pH < 7.1
  3. Neonatal cardiac resuscitation performed (includes CPAP, intubation and ventilation, or cardiopulmonary resuscitation)
  4. Neonatal encephalopathy (Severe brain injury diagnosed within the first 7 days of life defined as: was therapeutically cooled; and/or had decreased central tone or was comatose and had seizures of any kind; and/or had amplitude integrated electroencephalography (aEEG abnormality) in the first 24 hours of birth. )

CONTACTS AND LOCATIONS:
Overall Officials: Robert Rohling, PhD, Principal Investigator — The University of British Columbia
Locations (1):
- South Community Birth Program, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided